CLINICAL TRIAL: NCT00650793
Title: A Randomized, DB, PC and AC, Parallel Group, Dose-Response Study to Evaluate the Efficacy and Safety of 3 Fixed Dosages of Extended Release OROS� Paliperidone (6, 9, 12 mg/Day) and Olanzapine (10 mg/Day), With Open-Label Extension, in the Treatment of Subjects With Schizophrenia - Open Label Phase
Brief Title: A 52-week, Open-label Extension Study Following a 6-week, Double-blind, Placebo- and Active- Controlled Study (R076477-SCH-303) to Evaluate the Safety and Tolerability of Paliperidone ER in Subjects With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003376
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; paliperidone
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Extended Release OROS® Paliperidone

SUMMARY:
The purpose of the study was an Open Label Extension to a completed study that evaluated the efficacy and safety of 3 fixed dosages of Extended Release OROSÂ® Paliperidone

DETAILED DESCRIPTION:
This 52-week, open-label extension study followed a 6-week, double-blind, placebo- and active-controlled study (R076477-SCH-303) and was conducted at 52 sites in 11 countries. The primary objective of the open-label extension was the long-term assessment of safety and tolerability of flexibly-dosed ER OROS® paliperidone. The secondary objective was the assessment of long-term efficacy expressed as a function of change in the total Positive and Negative Syndrome Scale (PANSS) score, effect on positive and negative symptoms of schizophrenia by means of change in PANSS factor scores, and personal and social functioning, overall functioning, and quality of life parameters as measured by Personal and Social Performance Scale (PSP), Clinical Global Impression Scale - Severity (CGI-S), and Schizophrenia Quality of Life Scale (SQLS), respectively. Subjects in the open-label phase received flexibly dosed ER OROS® paliperidone (3 mg to 12 mg/day) for 52 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had completed the double-blind phase or discontinued due to lack of efficacy after at least 21 days of treatment, who signed the informed consent for the open-label phase, and who the investigator agreed that open-label treatment was in the best interest of the subject, were eligible to participate in the open-label phase.

Exclusion Criteria:

* Not eligible to enter the open-label phase if believed to be at significant risk for suicidal or violent behavior during the open-label extension trial, were pregnant, or had received an injection of a depot antipsychotic since entry into the preceding double-blind phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2004-03; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Long-term assessment of safety and tolerability of flexibly-dosed ER OROS® paliperidone.

SECONDARY OUTCOMES:
Assessment of long-term efficacy; Effect on positive and negative symptoms of schizophrenia; Personal and social functioning; Overall functioning; Quality of life parameters

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Kozma C, Dirani R, Canuso C, Mao L. Change in employment status over 52 weeks in patients with schizophrenia: an observational study. Curr Med Res Opin. 2011 Feb;27(2):327-33. doi: 10.1185/03007995.2010.541431. Epub 2010 Dec 15. PMID 21155708
- See also: A 52-week, open-label extension study following a 6-week, double-blind, placebo- and active- controlled study (R076477-SCH-303) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=524&filename=CR003376_CSR.pdf